CLINICAL TRIAL: NCT06531382
Title: Nurses Attitudes Towards Addressing Sexual Health - a Danish Crossectional Study
Brief Title: Danish Nurses Attitudes Towards Addressing Sexual Health
Status: Recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Kristina Holmegaard Nørskov, Post.doc. researcher, Rigshospitalet, Denmark
Other Study IDs: SIG seksualitet
Record Dates: First submitted 2024-07-10; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Sexuality; Communication; Sexual Dysfunction
MeSH Terms: conditions — Sexuality; Communication; Sexual Dysfunction, Physiological

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Nurses attitudes toward adressing sexual health in patients with cancer — Health professionals, within the field of cancer, attitude towards addressing sexual health with patients is unknown.
  The aim is to investigate the attitudes of Danish cancer nurses towards addressing sexual health in their clinical work, as well as to assess differences in perceived competences and knowledge.
  Method: The questionnaire Health professionals Attitudes towards Sexual Health-Danish version (PA-SH-D) is sent out to Danish cancer nurses via the Professional Society for Cancer Nurses. The questionnaire is sent out via a link via the RedCap database.
  The questionnaire link is sent out to members of the Professional Association for Cancer Nurses under the Danish Nursing Council, and it is sent out via their membership register.

SUMMARY:
Health professionals, within the field of cancer, attitude towards addressing sexual health with patients is unknown.

The aim is to investigate the attitudes of Danish cancer nurses towards addressing sexual health in their clinical work, as well as to assess differences in perceived competences and knowledge.

Method: The questionnaire Health professionals Attitudes towards Sexual Health-Danish version (PA-SH-D) is sent out to Danish cancer nurses via the Professional Society for Cancer Nurses. The questionnaire is sent out via a link via the RedCap database.

The questionnaire link is sent out to members of the Professional Association for Cancer Nurses under the Danish Nursing Council, and it is sent out via their membership register.

DETAILED DESCRIPTION:
Health professionals, within the field of cancer, attitude towards addressing sexual health with patients is unknown.

The aim is to investigate the attitudes of Danish cancer nurses towards addressing sexual health in their clinical work, as well as to assess differences in perceived competences and knowledge.

Method: The questionnaire Health professionals Attitudes towards Sexual Health-Danish version (PA-SH-D) is sent out to Danish cancer nurses via the Professional Society for Cancer Nurses. The questionnaire is sent out via a link via the RedCap database.

The questionnaire link is sent out to members of the Professional Association for Cancer Nurses under the Danish Nursing Council, and it is sent out via their membership register.

ELIGIBILITY:
Inclusion Criteria:

* Nurses working within the area of onkology or hematology in a danish hosptial or primary sector
* nurses having daily contact with patients with a cancer diagnosis

Exclusion Criteria:

* nurses not having daily contact with patients
* nurses not working within hematology or oncology

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: nurses
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Attitudes toward adressing sexual health | July 2024
  The main outcome measures Danish nurses attitudes toward addressing sexual health in their future professions, and differences in perceived competences and preparedness depending on the professional program.
  The measure is a Validated Questionnaire "health care students' attitudes towards addressing sexual health" (PA-SH-D).

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Østerbro, Denmark

IPD SHARING:
Plan to Share IPD: No